CLINICAL TRIAL: NCT04631796
Title: Clinical Characterization of an Investigational Soft Silicone Hydrogel Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLY935-E006
Record Dates: First submitted 2020-11-11; First posted 2020-11-17 (Actual); Results first posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Refractive Errors
Keywords: Vision; Contact lenses
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- LID020098 (Experimental): Lehfilcon A contact lenses worn in both eyes for 2 weeks. Lenses will be removed nightly for cleaning and disinfection.
  Interventions: Device: Lehfilcon A contact lenses; Device: Multipurpose disinfection solution

INTERVENTIONS:
Device: Lehfilcon A contact lenses — Silicone hydrogel contact lenses with investigational coating
  Other Names: LID020098
Device: Multipurpose disinfection solution — Solution for cleaning, disinfecting, and reconditioning silicone hydrogel contact lenses
  Other Names: OPTI-FREE® RepleniSH®

SUMMARY:
The primary objective of this study is to evaluate the overall clinical performance of an investigational silicone hydrogel contact lens over 2 weeks of daily wear.

DETAILED DESCRIPTION:
Participants will attend a Screening visit, a Dispense visit (0 to 4 days later), and a follow-up visit approximately 2 weeks after the Dispense visit.

ELIGIBILITY:
Inclusion Criteria:

* Understand and sign an Informed Consent that has been approved by an Institutional Review Board.
* Successful wear of spherical weekly/monthly soft contact lenses in both eyes for a minimum of 5 days per week and 8 hours per day during the past 3 months.
* Willing to stop wearing habitual contact lenses for the duration of study participation.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any condition that contraindicates contact lens wear, as determined by the Investigator.
* Any use of systemic or ocular medications that contraindicates contact lens wear, as determined by the Investigator.
* History of refractive surgery or plan to have refractive surgery during the study.
* Current or history of dry eye in either eye that, in the opinion of the Investigator, would preclude contact lens wear.
* Habitual contact lenses worn in an extended wear modality (routinely sleeping in lenses for at least 1 night per week) over the last 3 months prior to enrollment.
* Any use of topical ocular medications or artificial tear or rewetting drops that would require instillation during contact lens wear.
* Monovision or multifocal contact lens wear.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Trial Lead, CDMA Vision Care, Study Director — Alcon Research
Locations (3):
- United States (3):
  - Alcon Investigative Site, Orlando, Florida
  - Alcon Investigative Site, Bloomington, Illinois
  - Alcon Investigative Site, Powell, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 3 investigative sites located in the United States.
Pre-assignment Details: Of the 36 enrolled, 1 subject was exited from the study prior to product exposure as a screen failure. This reporting group includes all subjects/eyes exposed to any study lenses evaluated in this study, except for the lenses used with the purpose of power optimization (Safety Analysis Set).
Units Other Than Participants: eyes
Groups:
- LID020098: Lehfilcon A contact lenses worn in both eyes for 2 weeks. Lenses were removed nightly for cleaning and disinfection.
Period: Overall Study
Arm/Group | LID020098
Started | 35; 70 eyes
Completed | 35; 70 eyes
Not Completed | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Arm/Group | LID020098
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.4 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Front Surface Wettability, by Category
Description: Front surface wettability (i.e., assessment of the disruption of the front surface wettability of the contact lens) was assessed by the investigator for each eye individually. Front surface wettability was collected on a 5-point scale, where where Grade 0 = a smooth uniformly reflecting surface and Grade 4 = non-wettable lens surface. No formal hypothesis was predefined for the primary endpoint. No inferential testing was performed.
Time Frame: Dispense; Week 2 Follow-up
Population: Safety Analysis Set
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | LID020098
Number analyzed (Participants) | 35
Number analyzed (eyes) | 70
eyes
  Dispense, Grade 0 | 70
  Dispense, Grade 1 | 0
  Dispense, Grade 2 | 0
  Dispense, Grade 3 | 0
  Dispense, Grade 4 | 0
  Week 2 Follow-up, Grade 0 | 70
  Week 2 Follow-up, Grade 1 | 0
  Week 2 Follow-up, Grade 2 | 0
  Week 2 Follow-up, Grade 3 | 0
  Week 2 Follow-up, Grade 4 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AE's) were collected from time of consent to study exit, approximately 2 weeks.
Description: AE's were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of participants. This analysis population includes all subjects/eyes exposed to any study lenses evaluated in this study, except for the lenses used with the purpose of power optimization.
Groups:
- Pretreatment: Events reported in this group occurred prior to exposure to the study contact lenses
- LID020098 Ocular; LID020098 Nonocular: Events reported in this group occurred while exposed to the study contact lenses
Arm/Group | Pretreatment | LID020098 Ocular | LID020098 Nonocular
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/70 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/70 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/70 | 2/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=35) | LID020098 Ocular (N=70) | LID020098 Nonocular (N=35)
COVID-19 (Infections and infestations) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/96/NCT04631796/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/96/NCT04631796/SAP_001.pdf